CLINICAL TRIAL: NCT03170648
Title: Ear Acupuncture During Chemotherapy Infusion for Breast Cancer, a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Weidong Lu, MB, MPH, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-065
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Acupuncture; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Acupuncture (Experimental): Patients will receive a 30-minute session of a standardized ear acupuncture treatment Acupuncture needles will be gently manipulated to increase stimulation For each ear acupuncture session, the patient will have ear acupuncture therapy administered to each ear
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture has been studied in clinical trials in cancer patients and has been shown to be helpful for management of pain, nerve damage from chemotherapy, and nausea

SUMMARY:
This research study is evaluating ear acupuncture as a possible treatment to reduce symptoms related to receiving chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy drugs used to treat cancer can cause many symptoms. Some of the most common symptoms of receiving chemotherapy are nausea, vomiting, and anxiety. These symptoms can affect the quality of life of cancer patients. Medications can help ease these, but many patients continue to experience symptoms despite these treatments.

Acupuncture has been studied in clinical trials in cancer patients and has been shown to be helpful for management of pain, nerve damage from chemotherapy, and nausea.

Ear acupuncture is a type of acupuncture that involves the stimulation of points on the external ear. A few studies have suggested that ear acupuncture may help to reduce symptoms of nausea and anxiety during chemotherapy.

This study is being done to evaluate the potential benefits of using ear acupuncture to reduce symptoms like nausea and anxiety for women receiving chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically or cytologically proven Stage I-III breast cancer receiving intravenous chemotherapy on an every 14 days or every 21 days schedule
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Signed informed consent

Exclusion Criteria:

* Receiving weekly chemotherapy
* Unstable cardiac disease or myocardial infarction within 6 months prior to study entry
* Uncontrolled seizure disorder
* Pregnancy or potential pregnancy
* Active clinically significant uncontrolled infection
* Prior use of acupuncture within 3 months prior to the study entry
* Uncontrolled major psychiatric disorders, such as major depression or psychosis
* Metastatic breast or other cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Lu, MB, MPH, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang E, Lu W, Giobbie-Hurder A, Shin IH, Chen WY, Block CC, Partridge A, Jeselsohn RM, Tolaney SM, Freedman RA, Ligibel JA. Auricular Acupuncture During Chemotherapy Infusion in Breast Cancer Patients: A Feasibility Study. J Integr Complement Med. 2022 May;28(5):427-435. doi: 10.1089/jicm.2021.0256. Epub 2022 Mar 2. PMID 35238615
- See also: PubMed link — https://pubmed.ncbi.nlm.nih.gov/35238615/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 26 patients. Each patient is as its own control with education (cycle 2 of treatment) vs. the acupuncture (cycle 3 and 4 of treatment).
Groups:
- All Participants: During the first cycle of chemotherapy after study enrollment, participants (cycle 2 of treatment) were provided with an educational booklet developed by the National Cancer Institute. This booklet included information on chemotherapy, its side effects, and strategies for self-care.
  During the second and third cycles of chemotherapy after study enrollment (cycle 3 and 4 of treatment), the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
Period: Chemotherapy Education (Cycle 2)
Arm/Group | All Participants
Started | 26
Completed | 25
Not Completed | 1
Not completed — schedule conflict | 1
Period: Auricular Acupuncture (Cycle 3)
Arm/Group | All Participants
Started | 25
Completed | 24
Not Completed | 1
Not completed — Adverse Event | 1
Period: Auricular Acupuncture (Cycle 4)
Arm/Group | All Participants
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: During the first cycle of chemotherapy after study enrollment (cycle 2 of treatment), participants were provided with an educational booklet developed by the National Cancer Institute. This booklet included information on chemotherapy, its side effects, and strategies for self-care.
  During the second and third cycles of chemotherapy after study enrollment (cycle 3 and 4 of treatment), the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
ESAS-R Total Score [Mean (Standard Deviation); unit: units on a scale] — Edmonton Symptom Assessment System-Revised (ESAS-R) is a simple, 9-item scale that has been validated for assessing self-reported severity of common symptoms in cancer populations, and was used to evaluate symptom burden in this study. There are 9 symptoms included in this questionnaire: pain, fatigue, drowsiness, nausea, loss of appetite, shortness of breath, depression, anxiety, and lack of well-being. Each symptom is scored from 0 to 10 on a 11-point numerical rating scale. The total score ranges from 0 to 90, with higher scores indicating greater symptom burden.
  units on a scale | 7.4 (13.1)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Patient Enrollment and Intervention Adherence
Description: Feasibility was measured by:
  Enrollment of at least 20 patients (80% of the target sample size) within 3 months.
  Completion of at least 75% of scheduled auricular acupuncture sessions. Completion of at least 75% of ESAS assessments. Methods: Data were collected from patient enrollment logs, session attendance records, and ESAS assessment completion records.
Time Frame: Enrollment data over 3 months; Acupuncture attendance was recorded during Chemotherapy Cycles 2,3,4 ESAS were conducted at four time points for each cycle ESAS Assessments: Completion will were recorded up to 5 days post-infusion for Cycle 2-4
Measure: Number; unit: percentage of participants
Groups:
- All Participants: During the first cycle of chemotherapy after study enrollment (cycle 2 of treatment), participants were provided with an educational booklet developed by the National Cancer Institute. This booklet included information on chemotherapy, its side effects, and strategies for self-care.
  During the second and third cycles of chemotherapy (cycle 3 and 4 of treatment) after study enrollment, the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
Arm/Group | All Participants
Number analyzed (Participants) | 26
percentage of participants
  Percentage of target sample size | 100
  Percentage of participants completed auricular acupuncture sessions | 92.3
  Percentage of participants complete ESAS assessments | 84.6

2. Secondary Outcome: Changes in Edmonton Symptom Assessment System Revised (ESAS-R) Score Relative to Baseline at Education Cycle (Cycle 2)
Description: The Edmonton Symptom Assessment System-Revised Version (ESAS-R) is a 9-item scale that assesses the current severity of common symptoms. The ESAS-R has been validated in cancer populations. Each symptom is scored from 0 to 10 on an 11-point numerical rating scale, with total scores ranging from 0 to 90. Higher scores indicate a greater symptom burden.
Time Frame: Assessed at pre-education on day 1 (T1), post-education on day 1 (T2), day 2 (T3), day 5 (T4) of cycle 2 (Education)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: During the first cycle of chemotherapy after study enrollment (cycle 2 of treatment), participants were provided with an educational booklet developed by the National Cancer Institute. This booklet included information on chemotherapy, its side effects, and strategies for self-care.
  During the second and third cycles of chemotherapy after study enrollment (cycle 2 and 3 of treatment), the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
Arm/Group | All Participants
Number analyzed (Participants) | 24
score on a scale
  T2 vs. T1 | -1.1 (4.6)
  T3 vs. T1 | 1.4 (15.2)
  T4 vs. T1 | 7.4 (13.1)

3. Secondary Outcome: Changes in Edmonton Symptom Assessment System Revised (ESAS-R) Score Relative to Baseline at Acupuncture Cycle (Cycle 3 and Cycle 4)
Description: Scores of cycle 3 and cycle 4 are averaged. The Edmonton Symptom Assessment System-Revised Version (ESAS-R) is a 9-item scale that assesses the current severity of common symptoms. The ESAS-R has been validated in cancer populations. Each symptom is scored from 0 to 10 on an 11-point numerical rating scale, with total scores ranging from 0 to 90. Higher scores indicate a greater symptom burden.
Time Frame: Assessed at pre-acupuncture on day 1 (T1), post-acupuncture on day 1 (T2), day 2 (T3), day 5 (T4) of cycle 3 and cycle 4 (Acupuncture Cycles). Participants were followed up to 12 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: During the first cycle of chemotherapy after study enrollment (cycle 2 of the treatment), participants were provided with an educational booklet developed by the National Cancer Institute. This booklet included information on chemotherapy, its side effects, and strategies for self-care.
  During the second and third cycles of chemotherapy after study enrollment (cycle 3 and cycle 4 of the treatment), the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
Arm/Group | All Participants
Number analyzed (Participants) | 24
score on a scale
  T1 | 17.3 (12.3)
  T2 (post) vs. T1 (pre) | -3.0 (5.6)
  T3 (day 2) vs. T1 (pre) | -2.3 (10.2)
  T4 (day 5) vs. T1 (pre) | -0.5 (9.9)

4. Secondary Outcome: Changes in State-Trait Anxiety Inventory (STAI) Score Relative to Baseline Between Education (Cycle 2) and Acupuncture (Cycle 3 and 4)
Description: State-Trait Anxiety Inventory-State (STAI-S) is a validated and commonly used measure for evaluating a patient's current state of anxiety. It has been widely used in cancer populations. It consists of 20 items, with each item scored from 1 to 4, and the total score ranges from 20 to 80. Higher scores indicate a greater level of anxiety.
Time Frame: STAI were collected at four time points for each of the three cycles: 1) On the day of chemotherapy infusion or day 1, pre-education/acupuncture (T1); 2) Day 1, immediate post-education/acupuncture (T2); 3) Day 2 (T3); 4) Day 5 follow-up (T4)
Population: Patient-reported outcomes (ESAS-R, STAI-S, and MAT scores) during cycles 3 and 4 (acupuncture cycles) at each time point were averaged and compared with outcomes from cycle 2 (education cycle) using paired t-tests. The change from T1 to T2 is reported below.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 24
score on a scale
  T1 (pre) Cycle 2 (Education cycle) | 37.9 (11.0)
  T1 (pre): Cycle 3&4 (Acupuncture cycles) | 35.6 (11.8)
  T2 (post) vs. T1 (pre): cycle 2 (Education cycle) | -1.5 (4.3)
  T2 (post) vs. T1 (pre): Cycle 3&4 (Acupuncture cycles) | -4.9 (5.0)
  T3 (day 2) vs. T1 (pre): Cycle 2 (Education cycle) | 0.0 (9.3)
  T3 (day 2) vs. T1 (pre): Cycle 3 &4 (Acupuncture cycles) | -2.6 (5.7)
  T4 (day 5) vs. T1 (pre): cycle 2 (Education cycle) | 5.5 (9.8)
  T4 (day 5) vs. T1 (pre): Cycle 3&4 (Acupuncture cycles) | 0.4 (6.2)
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.02, t-test, 2 sided — T2 (post) vs.T1(pre)

5. Secondary Outcome: Number of Participants Experienced Acupuncture-related Adverse Effects
Description: The National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.0 were used to collect safety data related to adverse events, including skin bruising, hematoma, pre- syncope, syncope, and nausea.
Time Frame: Participants were followed up to 12 weeks.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
participants | 0

ADVERSE EVENTS:
Time Frame: Participants were followed up to 12 weeks.
Description: No SAE were reported.
Groups:
- Cycle 2 (Education Cycle): During the second cycle of chemotherapy after study enrollment, participants were provided with an educational booklet developed by the National Cancer Institute. This booklet included information on chemotherapy, its side effects, and strategies for self-care.
- Cycle 3 (Acupuncture Cycles): During the third cycle of chemotherapy after study enrollment, the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
- Cycle 4 (Acupuncture Cycles): During the fourth cycle of chemotherapy after study enrollment, the same participants received a 30-minute standardized auricular acupuncture treatment during chemotherapy infusion.
Arm/Group | Cycle 2 (Education Cycle) | Cycle 3 (Acupuncture Cycles) | Cycle 4 (Acupuncture Cycles)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/24

LIMITATIONS AND CAVEATS:
This was a pilot feasibility study with a small sample size, so data pertaining to patient-reported outcomes should be considered preliminary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03170648/Prot_SAP_000.pdf